CLINICAL TRIAL: NCT05620394
Title: Study of the Geometry of the Immature Human Femur Before the Age of 3 Years From Data Measured on CT Scan
Acronym: GFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7714
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Femur Fracture, Childhood
Keywords: Femur Fracture, Childhood
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Childhood fractures are the second most common presentation of abuse. The target population for screening for these injuries is children under the age of three who are unable to express themselves about the circumstances of the trauma, hence the need to develop a validated model to predict the outcome of trauma as well as the origin of a fracture.

Few morphological data are available in the literature for the femur concerning the period of rapid growth between 0 and 3 years of age.

ELIGIBILITY:
Inclusion criteria:

* Minor patient who died before the age of 3 years
* Whole body CT imaging performed post mortem on judicial requisition in the framework of a forensic procedure
* Absence of refusal in the medical file by the holders of parental authority concerning the re-use of their child's data for the purposes of this research

Exclusion criteria:

* Refusal manifested in the medical record by parental authority holders regarding the reuse of their child's data for the purpose of this research,
* Femur not fully assessable on imaging acquisition

Max Age: 3 Years | Sex: All
Age Groups: Child
Study Population: Minor patient who died before the age of 3 years
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To retrospectively characterize the variations in femur morphology during growth in a target pediatric population aged 0 to 3 years | Files analysed retrospectively from January 01, 2015 to February 29, 2020 will be examined
  To retrospectively characterize the variations in femur morphology during growth in a target pediatric population aged 0 to 3 years with the aim of later developing a numerical model to study fracture mechanisms for forensic applications

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Légale et Toxicologie - CHU de Strasbourg - France, Strasbourg, France